CLINICAL TRIAL: NCT01672528
Title: A Multicentre, Prospective Observational Study to Develop, Evaluate and Validate Patient Reported Outcome Measures (PROMs) for Patients Treated With Cardiac Ablation for Symptomatic Cardiac Arrhythmias
Brief Title: Patient Reported Outcome Measures for Ablation of Cardiac Arrhythmias
Status: Completed | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: National Institute for Health and Clinical Excellence (Unknown); University Hospital Birmingham NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); University College, London (Other)
Responsible Party: Principal Investigator, Dr Grace Carolan-Rees, Director, Cardiff and Vale University Health Board
Other Study IDs: 12-CAD-5351; RRK 4429 (Other: Birmingham R&D); 6125 (Other: Newcastle R&D)
Record Dates: First submitted 2012-08-16; First posted 2012-08-27 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Cardiac Arrhythmia
Keywords: Patient Reported Outcome Measures; PROMs; Cardiac arrhythmia; Cardiac ablation
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac arrhythmia patients: Patients with cardiac arrhythmias consented to and awaiting a cardiac ablation procedure or post ablation.
  Interventions: Other: Interview; Other: Questionnaires

INTERVENTIONS:
Other: Interview — Patient participates in a face-to-face interview to facilitate development of the new disease specific questionnaire
  Other Names: Disease specific questionnaire; EQ5D5L
Other: Questionnaires — Patients will be sent questionnaires before their procedure, 8 - 12 after their procedure and at 1 and 5 years post procedure
  Other Names: Disease specific questionnaire; EQ5D

SUMMARY:
A multicentre, prospective observational study to develop, evaluate and validate Patient Reported Outcome Measures (PROMs) for patients treated with cardiac ablation for symptomatic cardiac arrhythmias

DETAILED DESCRIPTION:
This study aims to develop, evaluate and validate disease specific PROMs for patients in the UK treated with cardiac ablation for cardiac arrhythmias. The potential benefits include support for clinicians to improve their performance, assisting patients in making informed choices and strengthening audit and research.

Phase 1 of the study will involve patient interviews with approximately 30 patients from 2 sites. These, together with input from a multidisciplinary team, will aim to improve drafts of disease specific questionnaires. This will be followed by Phase 2 which will trial the questionnaires in a group of approximately 600 patients from three sites. In Phase 2 patients will be asked to complete a pre-procedure questionnaire relating to their symptoms, quality of life and procedure expectations. They will also be sent post-procedure questionnaires relating to procedural outcomes, symptoms and quality of life at 8-16 weeks post procedure and at 1 and 5 years post-procedure.

The responses obtained from these PROMs will be used to undertake recommended statistical tests of reliability and validity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic cardiac arrhythmias
* Consented to and awaiting a cardiac ablation procedure
* Able to read, write and understand English or Welsh
* Capable of giving informed written consent

Exclusion Criteria:

* Not able to read, write and understand English or Welsh
* Not able to provide informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac arrhythmia clinic
Sampling Method: Non-Probability Sample
Enrollment: 586 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Is a newly developed disease specific tool able to accurately detect changes in health status following ablation for symptomatic cardiac arrhythmias? | Up to 5 years post ablation
  This will be measured using responses to the new tool, EQ5D5L and clinical outcomes. Statistical evidence of the reliability and validity of the instruments will be illustrated via standard statistical methods.

SECONDARY OUTCOMES:
Do replies to the questionnaires show that the tool is responsive to change following ablation treatment? | Average 10 weeks post ablation
Do PROMs responses show concurrent, convergent and discriminant validity; corresponding with responses to EQ5D and clinical outcomes? | Up to 5 years post-ablation.
Is the tool sensitive to detecting whether patient expectations are met following ablation procedures for cardiac arrhythmias? | Average 10 weeks post ablation

CONTACTS AND LOCATIONS:
Overall Officials: Grace Carolan-Rees, PhD, Principal Investigator — Cardiff and Vale University Health Board
Locations (3):
- United Kingdom (3):
  - University Hospitals Birmingham Foundation Trust, Birmingham
  - Cardiff and Vale University Health Board, Cardiff
  - Newcastle Upon Tyne Hospitals NHS Trusts, Newcastle

REFERENCES:
- [Derived] Withers KL, Wood KA, Carolan-Rees G, Patrick H, Lencioni M, Griffith M. Living on a knife edge-the daily struggle of coping with symptomatic cardiac arrhythmias. Health Qual Life Outcomes. 2015 Jun 24;13:86. doi: 10.1186/s12955-015-0282-9. PMID 26104746